CLINICAL TRIAL: NCT05508932
Title: Atrial Fibrillation in Beta-Thalassemia
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Matteo Bertini, Associate Professor, University Hospital of Ferrara
Other Study IDs: 419/2022/Oss/AOUFe
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Atrial Fibrillation; Thalassemia
Keywords: Atrial Fibrillation; Thalassemia; Thalassaemia; Arrhythmia; Hemoglobinopathies
MeSH Terms: conditions — Atrial Fibrillation; Thalassemia; Arrhythmias, Cardiac; Hemoglobinopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Beta-thalassemia: Patients with Beta-thalassemia undergoing a cardiological evaluation

SUMMARY:
The study aims to evaluate the clinical, laboratory and instrumental differences that exist between beta-thalassemia patients with atrial fibrillation and those not affected by arrhythmia.

DETAILED DESCRIPTION:
Observational, retrospective and prospective, single-center study, which involves the collection of clinical, laboratory, electrocardiographic and imaging data of patients with major or intermediate thalassemia who have performed, from 2012 to 2022, or will perform in the next 10 years, a cardiological evaluation at the Cardiology Unit of the University Hospital of Ferrara. Patients will be divided into two groups: thalassemia patients with atrial fibrillation (paroxysmal, persistent or permanent) and thalassemia patients with no history of atrial fibrillation.

The objective of the study is to evaluate whether there is a different prevalence of the characteristics analyzed among these patient populations.

As secondary outcome, the effect of SGLT2-inhibitors (empaglifozin, dapaglifozin, ...) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Transfusion-dependent Beta-thalassemia;
2. Follow-Up at the Cardiology Unit of the University Hospital of Ferrara;
3. Electrocardiogram performed;
4. Echocardiogram performed.

Exclusion Criteria:

1. Age <18 years;
2. State Of pregnancy;
3. Inability to give informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Transfusion-dependent Beta-thalassemia patients
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2032-06-01 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Atrial fibrillation | 10 years
  New onset of Atrial Fibrillation documented at ECG

SECONDARY OUTCOMES:
Thromboembolism | 10 years
  Stroke or peripheral embolization
Epicardial adipose tissue | Baseline
  Thickness of fat depot in epicardial region
SGLT2 effect on Hb | 6 months
  rise in hemoblogin levels

CONTACTS AND LOCATIONS:
Locations (1):
- Matteo Bertini, Ferrara, Italy

REFERENCES:
- [Derived] Malagu M, Marchini F, Longo F, Zuin M, Orazio G, Capanni A, Berloni ML, Frascaro F, Tonet E, Cossu A, Culcasi M, Bonsi B, Balla C, Vitali F, Bertini M. Association between epicardial adipose tissue and transfusion-dependent beta-thalassemia. Int J Cardiovasc Imaging. 2025 Nov;41(11):2255-2263. doi: 10.1007/s10554-025-03535-2. Epub 2025 Oct 9. PMID 41065927